CLINICAL TRIAL: NCT05890469
Title: Effect of Implant Surface Material and Topography on Bone Regeneration: A Two-centre, Parallel-group, Pilot Study
Brief Title: Effect of Implant Surface Material and Topography on Bone Regeneration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRAS:321927
Record Dates: First submitted 2023-04-12; First posted 2023-06-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant; Guided Bone Regeneration; Biomarkers; Saliva

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia surface implant and guided bone regeneration (Test) (Experimental): Zirconia surface implant (Straumann PURE®, Basel, Switzerland) and guided bone regeneration (GBR) with a porcine collagen membrane (Bio-Gide®, Geistlich, Wolhusen, Switzerland) and a deproteinized bovine bone substitute (Bio-Oss Collagen®, Geistlich, Wolhusen, Switzerland).
  Interventions: Combination Product: Zirconia surface implant and guided bone regeneration
- Hydrophilic titanium surface implant and guided bone regeneration (Control) (Other): Hydrophilic titanium surface implant (Straumann Standard Plus (SP) Tissue level, SLActive®, Basel, Switzerland) and guided bone regeneration (GBR) with a porcine collagen membrane (Bio-Gide®, Geistlich, Wolhusen, Switzerland) and a deproteinized bovine bone substitute (Bio-Oss Collagen®, Geistlich, Wolhusen, Switzerland).
  Interventions: Combination Product: Hydrophilic titanium surface implant and guided bone regeneration

INTERVENTIONS:
Combination Product: Zirconia surface implant and guided bone regeneration — The Straumann® PURE Ceramic Implant System is made from 100 % yttria-stabilized zirconia. Its surface features a topography characterized by macro- and micro-roughness to offer a structure for cell attachment and the osseointegration of this surface has been successfully proven. Owing to the increasing aesthetic standards in the field of implant dentistry and the concerns on sensitivity to titanium, there has been a growing interest towards metal-free implant rehabilitation.
  Guided bone regeneration (GBR) will be performed simultaneously with the implant placement with the aim to re-establish the bone contour. A bovine osteoconductive graft (Bio-Oss collagen®, Geistlich, Wolhusen, Switzerland) will be placed on the buccal aspect of the implant and covered with a collagen membrane (Bio-Gide®, Geistlich, Wolhusen, Switzerland).
  Arms: Zirconia surface implant and guided bone regeneration (Test)
Combination Product: Hydrophilic titanium surface implant and guided bone regeneration — The Straumann® Standard Plus (SP) Implant is a Soft Tissue Level Implant with a smooth neck section of 1.8 mm. It has a fundamentally improved hydrophilic surface chemistry (SLActive®) which accelerates the osseointegration process in the early healing phase.
  Guided bone regeneration (GBR) will be performed simultaneously with the implant placement with the aim to re-establish the bone contour. A bovine osteoconductive graft (Bio-Oss collagen®, Geistlich, Wolhusen, Switzerland) will be placed on the buccal aspect of the implant and covered with a collagen membrane (Bio-Gide®, Geistlich, Wolhusen, Switzerland).
  Arms: Hydrophilic titanium surface implant and guided bone regeneration (Control)

SUMMARY:
Dental implants have been on the market for several years and they are routinely used to replace single/multiple missing teeth with a high success rate. However, there is still a limited number of studies comparing hydrophilic titanium and zirconia implants. In addition, there is no data available on the signalling pathways and the expression of healing biomarkers involved in the early stages of osseointegration around zirconia surface implants placed with guided bone regeneration (GBR).

This study aims 1) to describe and compare the early wound healing molecular pathways, and the 2) vascularization patterns of mucosal tissues after the placement of hydrophilic titanium or zirconia implants with simultaneous guided bone regeneration (GBR).

In this study, the investigators will assess the expression of inflammatory, angiogenesis and osseous biomarkers of PICF at 3, 7, 15 and 30 days after the placement of hydrophilic titanium or zirconia dental implants with simultaneous GBR and of saliva at day 1, 3, 7, 15 and 30.

DETAILED DESCRIPTION:
This is a two-centre prospective, parallel-group pilot study which will consist of 10-11 visits over a minimum period of 14 months. The study will take place at the Centre for Oral Clinical Research (COCR), at the Institute of Dentistry, Barts and The London School of Medicine and Dentistry, Queen Mary University of London (main centre), United Kingdom and at Clinic of Reconstructive Dentistry, University of Zurich, Zurich in accordance with local guidelines and procedures/interventions detailed below.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 25 years old
* Good/controlled medical and psychological health
* Good oral hygiene (full mouth plaque scores [FMPS< 30%])
* Need of a single-tooth replacement in the aesthetic (incisor, canine or premolar) region
* At least one neighbouring natural tooth present
* A functional occlusion with a minimum of four occlusal units (i.e., pairs of occluding posterior teeth)
* At least 3 months of post-extraction socket healing had occurred in the edentulous site and no ridge preservation was performed
* After implant placement, presence of buccal bone dehiscence/fenestration or thin buccal bone plate (<2mm) requiring guided bone regeneration (GBR) (including contour augmentation) [to be confirmed after implant placement]
* Willingness to read and sign a copy of the Informed Consent Form (ICF) after reading the Patient Information Sheet (PIS), and after the nature of the study has been fully explained and potential questions fully answered

Exclusion Criteria:

* Any known systemic disease severely affecting bone metabolism (e.g., Cushing's syndrome, Crohn's disease, rheumatoid arthritis, osteoporosis or diabetes type I and uncontrolled diabetes type II)
* Self-reported HIV or viral hepatitis
* Self-reported alcoholism or chronic drug abuse
* Smokers (including current smokers or former smokers who had quit for < 3 months); patients reporting use of vape/ e-cigarettes will also be excluded
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing, which can affect interpretation of study results)
* Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status or bone metabolism (e.g., bisphosphonates, hormone replacement therapy, immunosuppressants) within 1 month before baseline visit
* Chronic treatment with anticoagulants (including aspirin), corticosteroids, immunosuppressants or other medications that may influence blood coagulation/count
* Antibiotic or anti-inflammatory therapy during the month preceding the baseline exam.
* Untreated caries lesions and untreated/uncontrolled periodontal disease. If patients require periodontal treatment (non-surgical and/or surgical), this will be arranged outside the study protocol and completed prior to enrolment
* Inadequate keratinized tissue width (<2 mm) in the mid-buccal aspect of the area to be treated in the study
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene in the area of implant placement
* Patients requiring maxillary sinus lift surgery before implant placement
* Self-reported bruxism
* Patients not willing to receive animal-derived biomaterials for GBR
* Patients suffering from a known psychological disorder or with limited mental capacity or language skills such that study information could not be understood, informed consent could not be obtained, or simple instructions could not be followed
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Changes in the expression of inflammatory, angiogenesis and osseous biomarkers of PICF and saliva | 1,3, 7, 15 and 30 days after the placement of hydrophilic titanium or zirconia dental implants.
  The expression of inflammatory, angiogenesis and osseous biomarkers of PICF at 3, 7, 15 and 30 days after the placement of hydrophilic titanium or zirconia dental implants with simultaneous GBR and of saliva at day 1, 3, 7, 15 and 30.

SECONDARY OUTCOMES:
Blood flow changes | immediately after, 1, 3, 7, 15 and 30 days after the placement of hydrophilic titanium or zirconia dental implants
  Blood flow changes immediately after, at 1, 3, 7, 15 and 30 days after implant placement (IP)
Soft tissue volume changes | immediately after,1, 3, 7, 15, 30 days and 3 months after IP, at loading and 6 months after implant loading
  Soft tissue volume changes immediately after, at 1, 3, 7, 15, 30 days and 3 months after IP, at loading and 6 months after implant loading
Peri-implant bone level | 6 months after implant loading
  Peri-implant bone level 6 months after loading, using CBCT images
Full mouth plaque score (FMPS) | 6 months after implant loading
  FMPS will be recorded as a percentage of total surfaces (6 sites per tooth/implant), which reveal the presence of plaque. A binary score will be assigned to each surface (1 for plaque present, 0 for absent).
Full mouth bleeding score (FMBS) | 6 months after implant loading
  FMBS will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of bleeding within 10 - 30 seconds following periodontal probing. A binary score will be assigned to each surface (1 for bleeding present, 0 for bleeding absent).
Probing pocket depth (PPD) | 6 months after implant loading
  PPD will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual)
Gingival recession (REC) | 6 months after implant loading
  REC will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual)
Clinical attachment level (CAL) | 6 months after implant loading
  CAL will be calculated considering the values for PPD and REC in mm
Suppuration | 6 months after implant loading
  Suppuration will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of suppuration following periodontal probing. A binary score will be assigned to each surface (1 for suppuration present, 0 for suppuration absent)
Patient satisfaction at 6 months after loading | 6 months after implant loading
  Patient satisfaction regarding the overall implant treatment using a subjective outcome questionnaire at 6 months post loading.
Changes in the pink esthetic score (PES) | 6 months after implant loading
  Changes in the pink esthetic score (PES) from loading to 6 months after loading
Changes in the white esthetic score (WES) | 6 months after implant loading
  Changes in the white esthetic score (WES) from loading to 6 months after loading
Changes in the papilla fill index (PFI) | 6 months after implant loading
  Changes in the papilla fill index (PFI) from loading to 6 months after loading

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, Principal Investigator — QMUL
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust Dental Hospital, London
  - Centre for Oral Clinical Research, London